CLINICAL TRIAL: NCT00887094
Title: Acute and Subacute Effects of Aerobic Training vs Aerobic/Resistance Training Upon Glucose Profile Evaluated Through Continuous Glucose Monitoring System in Type 2 Diabetes
Brief Title: Aerobic Training, Aerobic-resistance Training and Glucose Profile (CGMS) in Type 2 Diabetes
Acronym: CGMSexercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Dr. Beatriz Schaan, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-180
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Type 2; Treatment; Exercise
Keywords: Diabetes mellitus; Exercise; Endurance; Resistance; Continuous glucose monitoring system
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Experimental): One bout of aerobic physical training will be performed on a cycle ergometer for 50 min
  Interventions: Behavioral: Acute aerobic exercise
- Aerobic-resistance exercise (Experimental): One bout of aerobic-resistance physical training will be performed on a cycle ergometer added by a strenght training for 50 min (total)
  Interventions: Behavioral: Acute aerobic-resistance exercise

INTERVENTIONS:
Behavioral: Acute aerobic exercise — Aerobic exercise (on a cycle ergometer, for 50 min)
  Other Names: There are no other names
  Arms: Aerobic exercise
Behavioral: Acute aerobic-resistance exercise — Aerobic-resistance exercise (on a cycle ergometer plus strength training, for 50 min in total)
  Other Names: There are no other names
  Arms: Aerobic-resistance exercise

SUMMARY:
Many studies were already performed showing beneficial cardiovascular and metabolic effects of physical training for type 2 diabetic patients. However, glucose profile during and immediately after a short period of aerobic and/or resistance training was not studied yet. Continuous glucose monitoring system (CGMS) has now been added to the repertoire of technological devices useful in the management of patients with diabetes. Such monitoring enables clinicians to detect occult hypoglycemia and hyperglycemia not otherwise discernable with intermittent testing of blood glucose. The main aim of the present study is to investigate continuous blood glucose profile (using CGMS) over 72h, beginning 24h before and ending 24h after a single bout of aerobic or aerobic/resistance physical training in type 2 diabetic patients.

DETAILED DESCRIPTION:
Many studies were already performed showing beneficial cardiovascular and metabolic effects of physical training for type 2 diabetic patients. However, glucose profile during and immediately after a short period of aerobic and/or resistance training was not studied yet. Continuous glucose monitoring system (CGMS) has now been added to the repertoire of technological devices useful in the management of patients with diabetes. Such monitoring enables clinicians to detect occult hypoglycemia and hyperglycemia not otherwise discernable with intermittent testing of blood glucose. The main aim of the present study is to investigate continuous blood glucose profile (using CGMS) over 72h, beginning 24h before and ending 24h after a single bout of aerobic or aerobic/resistance physical training in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients treated with diet and metformin, 35-65 years old

Exclusion Criteria:

* Type 1 diabetic patients
* Treatment with insulin or sulphonylureas or glitazones
* Proliferative retinopathy
* Severe autonomic neuropathy
* Coronary artery disease
* Baseline fasting plasma glucose>200 mg/dl
* Peripheral artery disease
* Amputation
* Heart failure
* Diabetic nephropathy
* Renal failure

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Reduction of the prevalence of hyperglycemic peaks during a 24-h period after a bout of aerobic or aerobic/resistance exercise in type 2 diabetes patients on metformin/diet therapy. | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Schaan, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Figueira FR, Umpierre D, Casali KR, Tetelbom PS, Henn NT, Ribeiro JP, Schaan BD. Aerobic and combined exercise sessions reduce glucose variability in type 2 diabetes: crossover randomized trial. PLoS One. 2013;8(3):e57733. doi: 10.1371/journal.pone.0057733. Epub 2013 Mar 11. PMID 23536769
- [Derived] Figueira FR, Umpierre D, Ribeiro JP, Tetelbom PS, Henn NT, Esteves JF, Schaan BD. Accuracy of continuous glucose monitoring system during exercise in type 2 diabetes. Diabetes Res Clin Pract. 2012 Dec;98(3):e36-9. doi: 10.1016/j.diabres.2012.09.033. Epub 2012 Oct 4. PMID 23041227